CLINICAL TRIAL: NCT06595082
Title: Evaluation of the Consumption of Lupins in Brine on Metabolic Markers in Healthy Individuals
Acronym: SUPERLUPINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Teramo (Other)
Responsible Party: Principal Investigator, Mauro Serafini, Professor, University of Teramo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Superlupino
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lipid Disorder; Systemic Inflammatory Response
Keywords: Lupins; Blood Lipids; Inflammation
MeSH Terms: conditions — Lipid Metabolism Disorders; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 grams Lupin (Active Comparator): 30 grams per week of lupins in brine
  Interventions: Dietary Supplement: 4-week lupins in brine consumption
- 600 grams Lupin and dietary suggestion (Experimental): 600 grams per week of lupins in brine and dietary suggestion of lowering of two servings per week among meat, processed meat and/or cheese.
  Interventions: Dietary Supplement: 4-week lupins in brine consumption and dietary suggestion

INTERVENTIONS:
Dietary Supplement: 4-week lupins in brine consumption — Volunteers were asked to consume lupins in brine for 4 weeks.
  Arms: 30 grams Lupin
Dietary Supplement: 4-week lupins in brine consumption and dietary suggestion — Volunteers were asked to consume lupins in brine for 4 weeks and refrain to two servings per week of meat or processed meat or cheese.
  Arms: 600 grams Lupin and dietary suggestion

SUMMARY:
The aim of the project was the evaluation of the effects of the consumption of different amounts of lupins in brine on lipid, glucose, inflammatory, oxidative stress, gut microbiota profile and (epi)genetic markers in healthy volunteers, by means of a 4-week 2-arm parallel randomized controlled trial.

DETAILED DESCRIPTION:
Epidemiological and intervention studies confirm a tight relationship between lifestyle - and particularly dietary choices - and human health. Among the dietary patterns, it has been showed that the adherence to a plant-based diet, i.e. Mediterranean diet, may have a pivotal role in promoting a health longevity and counteracting cardiovascular, neurological and cancer-related diseases. In fact, the abundant consumption of fruit, vegetables, cereals and pulses leads to a high intake of vegetable proteins, unsaturated fatty acids, minerals, vitamins, fibre and bioactive compounds which may have anti-inflammatory, antioxidant, anti-atherosclerotic, hypocholesterolemic and antimicrobial activities. In particular, there is a growing interest for valorization of pulses, among which lupins represent a good alternative as healthy snack but also as serving to be used during the principal meal. Lupins are traditional legumes of the Mediterranean basin, and they represent a good source of bioactive peptides, soluble fibre and minerals. Different trials evaluated the health effects of the consumption lupin derived products in humans concluding that it may lead to a decrease of blood pressure, reduction of blood glucose, cholesterol, triglycerides and uric acid.

Nevertheless, there is still a lack of information regarding the effects of the consumption of whole lupins, and in particular in one of the most sold forms, as in brine.

In this parallel randomized controlled trial, 60 healthy volunteers were randomly allocated for a 4-week consumption of:

* Active comparator arm: 30 grams per week of lupins in brine;
* Experimental arm: 600 grams per week of lupins in brine and the suggestion of reduction of at least two servings per week of meat, processed meat and/or cheese;

At baseline and after 4 weeks of dietary intervention, subjects were visited in medical facility and asked to provide blood, urine, saliva, feces for the evaluation of:

* Anthropometric and blood pressure parameters;
* Blood lipid and carbohydrate profile;
* Blood transaminase parameters;
* Blood and urine inflammation markers;
* Leucocyte and saliva DNA genetic and epigenetic markers;
* Fecal profile of gut microbiota. In addition, volunteers filled in different questionnaires regarding their dietary habits, the physical activity and the gut healthiness.

ELIGIBILITY:
Inclusion Criteria:

* BMI included between 18.5 and 29.9 kg/m2;
* Omnivorous diet;
* Consumption of more than 6 servings of meat, processed meat and/or cheese;

Exclusion Criteria:

* Antibiotic treatment within 3 months prior the dietary intervention;
* Chronic diseases
* Surgeries
* Dieting
* Pregnant or lactating

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Variation of plasma lipids | 4 weeks
  Measure of plasma concentrations (mg/dL) of triglycerides before and after dietary intervention.
  Statistical analysis of the primary outcome was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.

SECONDARY OUTCOMES:
Variation of anthropometric parameters | 4 weeks
  Measure of body weight (kg), height (m), BMI (kg/m2) fat mass (kg), free fat mass (kg) before and after dietary intervention. Weight (in kilograms) and height (and in meters) will be combined to report BMI in kg/m^2).
  Statistical analysis of the secondary outcome was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of blood pressure parameters | 4 weeks
  Measure of blood pressure (mmHg).
  Statistical analysis of the secondary outcome was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of blood glucose | 4 weeks
  Measure of blood glucose (mg/dL) before and after dietary intervention.
  Statistical analysis of the secondary outcomes was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of blood insulin | 4 weeks
  Measure of blood insulin (µUI/mL) before and after dietary intervention.
  Statistical analysis of the secondary outcomes was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of C-peptide | 4 weeks
  Measure of blood C-peptide (ng/mL) before and after dietary intervention.
  Statistical analysis of the secondary outcomes was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of blood lipid-related parameters | 4 weeks
  Measure of blood total (mg/dL), LDL- (mg/dL), HDL- (mg/dL) cholesterol before and after dietary intervention.
  Statistical analysis of the secondary outcomes was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of transaminase parameters | 4 weeks
  Measure of blood aspartate transaminase (AST, U/L), alanine transaminase (ALT, U/L), γ-glutamyltransferase (GGT, U/L )before and after dietary intervention.
  Statistical analysis of the secondary outcomes was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of inflammatory parameters | 4 weeks
  Measure of blood C-reactive protein (CRP, mg/dL) and uric acid (mg/dL) before and after dietary intervention.
  Statistical analysis of the secondary outcomes was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of citokine and interleukine parameters | 4 weeks
  Measure of blood interleukins (IL) IL-1β, IL-4, IL-6, IL-10, IL-17, IL-18, interferon-γ, tumor necrosis factor-α (pg/mL) before and after dietary intervention.
  Statistical analysis of the secondary outcomes was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of urinary inflammatory parameters | 4 weeks
  Measure of urinary 8-isoprotaglandin F2α (8-iso-PGF2α, ng/mL) before and after dietary intervention before and after dietary intervention.
  Statistical analysis of the secondary outcomes was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of genetic and epigenetic expression of inflammatory mediators parameters | 4 weeks
  Measure of DNA methylation on CpG sites from peripheral blood mononuclear cell (PBMC) cells (% on single site) and expression of miRNA on saliva samples (fold change over control) before and after dietary intervention.
  Statistical analysis of the secondary outcomes was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.
Variation of gut microbiota profile parameters | 4 weeks
  Measure of fecal microbiota composition (colony-forming unit, CFU/g) and short chain fatty acids (SCFA) before and after dietary intervention.
  Statistical analysis of the secondary outcomes was performed within and between each single intervention-arm. Further, a post-hoc subdivision of the study participants by means of anthropometrics or metabolic marker cut-off value was applied, and statistical differences of the primary outcome have been considered.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Serafini, PhD, Principal Investigator — University of Teramo; Donato Angelino, PhD, Study Director — University of Teramo
Locations (1):
- University of Teramo, Teramo, Italy

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and datasets analysed during the current study are available from the Principal Investigator on reasonable request prior email contact.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data are available since the end of the intervention study for a 1-year time frame.
Access Criteria: Contact to Principal Investigator

REFERENCES:
- [Background] Bahr M, Fechner A, Kramer J, Kiehntopf M, Jahreis G. Lupin protein positively affects plasma LDL cholesterol and LDL:HDL cholesterol ratio in hypercholesterolemic adults after four weeks of supplementation: a randomized, controlled crossover study. Nutr J. 2013 Aug 1;12:107. doi: 10.1186/1475-2891-12-107. PMID 23902673
- [Background] Bahr M, Fechner A, Kiehntopf M, Jahreis G. Consuming a mixed diet enriched with lupin protein beneficially affects plasma lipids in hypercholesterolemic subjects: a randomized controlled trial. Clin Nutr. 2015 Feb;34(1):7-14. doi: 10.1016/j.clnu.2014.03.008. Epub 2014 Apr 1. PMID 24746974
- [Background] Belski R, Mori TA, Puddey IB, Sipsas S, Woodman RJ, Ackland TR, Beilin LJ, Dove ER, Carlyon NB, Jayaseena V, Hodgson JM. Effects of lupin-enriched foods on body composition and cardiovascular disease risk factors: a 12-month randomized controlled weight loss trial. Int J Obes (Lond). 2011 Jun;35(6):810-9. doi: 10.1038/ijo.2010.213. Epub 2010 Oct 12. PMID 20938438
- [Background] D'Addario C, Pucci M, Bellia F, Girella A, Sabatucci A, Fanti F, Vismara M, Benatti B, Ferrara L, Fasciana F, Celebre L, Vigano C, Elli L, Sergi M, Maccarrone M, Buzzelli V, Trezza V, Dell'Osso B. Regulation of oxytocin receptor gene expression in obsessive-compulsive disorder: a possible role for the microbiota-host epigenetic axis. Clin Epigenetics. 2022 Mar 31;14(1):47. doi: 10.1186/s13148-022-01264-0. PMID 35361281
- [Background] D'Addario C, Pucci M. DNA Methylation Analysis of Cnr1 Gene Promoter. Methods Mol Biol. 2023;2576:373-384. doi: 10.1007/978-1-0716-2728-0_31. PMID 36152203
- [Background] Fanti F, Vincenti F, Montesano C, Serafini M, Compagnone D, Sergi M. dLLME-muSPE extraction coupled to HPLC-ESI-MS/MS for the determination of F2alpha-IsoPs in human urine. J Pharm Biomed Anal. 2020 Jul 15;186:113302. doi: 10.1016/j.jpba.2020.113302. Epub 2020 Apr 17. PMID 32353681
- [Background] Miglio C, Peluso I, Raguzzini A, Villano DV, Cesqui E, Catasta G, Toti E, Serafini M. Antioxidant and inflammatory response following high-fat meal consumption in overweight subjects. Eur J Nutr. 2013 Apr;52(3):1107-14. doi: 10.1007/s00394-012-0420-7. Epub 2012 Jul 19. PMID 22810465
- [Background] Partridge L, Deelen J, Slagboom PE. Facing up to the global challenges of ageing. Nature. 2018 Sep;561(7721):45-56. doi: 10.1038/s41586-018-0457-8. Epub 2018 Sep 5. PMID 30185958
- [Background] Peluso I, Miglio C, Morabito G, Ioannone F, Serafini M. Flavonoids and immune function in human: a systematic review. Crit Rev Food Sci Nutr. 2015;55(3):383-95. doi: 10.1080/10408398.2012.656770. PMID 24915384
- [Background] Peluso I, Villano DV, Roberts SA, Cesqui E, Raguzzini A, Borges G, Crozier A, Catasta G, Toti E, Serafini M. Consumption of mixed fruit-juice drink and vitamin C reduces postprandial stress induced by a high fat meal in healthy overweight subjects. Curr Pharm Des. 2014;20(6):1020-4. doi: 10.2174/138161282006140220144802. PMID 23701571
- [Background] Ruscica M, Pavanello C, Gandini S, Gomaraschi M, Vitali C, Macchi C, Morlotti B, Aiello G, Bosisio R, Calabresi L, Arnoldi A, Sirtori CR, Magni P. Effect of soy on metabolic syndrome and cardiovascular risk factors: a randomized controlled trial. Eur J Nutr. 2018 Mar;57(2):499-511. doi: 10.1007/s00394-016-1333-7. Epub 2016 Oct 18. PMID 27757595
- [Background] Willett W, Rockstrom J, Loken B, Springmann M, Lang T, Vermeulen S, Garnett T, Tilman D, DeClerck F, Wood A, Jonell M, Clark M, Gordon LJ, Fanzo J, Hawkes C, Zurayk R, Rivera JA, De Vries W, Majele Sibanda L, Afshin A, Chaudhary A, Herrero M, Agustina R, Branca F, Lartey A, Fan S, Crona B, Fox E, Bignet V, Troell M, Lindahl T, Singh S, Cornell SE, Srinath Reddy K, Narain S, Nishtar S, Murray CJL. Food in the Anthropocene: the EAT-Lancet Commission on healthy diets from sustainable food systems. Lancet. 2019 Feb 2;393(10170):447-492. doi: 10.1016/S0140-6736(18)31788-4. Epub 2019 Jan 16. No abstract available. PMID 30660336
- [Background] Serafini M, Jirillo E. Mangiare per prevenire. L'Immunonutrizione a tavola. 2015. Books & Company Editore.
- [Background] Serafini M, Miglio C. Dietary plant products and human health. New evidences about the effects on degenerative diseases. 2011. Nova Science Publisher. NY